CLINICAL TRIAL: NCT03499951
Title: Remote Wheelchair Skills Training Efficacy Coordinating Center
Brief Title: Remote Wheelchair Skills Training Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Boninger, Professor and UPMC Endowed Vice Chair for Research, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO18010289
Record Dates: First submitted 2018-03-19; First posted 2018-04-17 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Spinal Cord Injuries
Keywords: Quality of life; Participation; Training
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wheelchair Skills Trainers (Other): Individuals will receive remotely delivered wheelchair skills training, after which they will be assessed on their ability to teach the Wheelchair Skills Trainees a series of wheelchair skills in a one-on-one environment. The intervention for this group is Wheelchair Skills Training - Remote.
  Interventions: Behavioral: Wheelchair Skills Training - Remote
- Wheelchair Skills Trainees (Other): Individuals will receive one-on-one wheelchair skills training from the Wheelchair Skills Trainers. The intervention for this group is Wheelchair Skills Training - In Person.
  Interventions: Behavioral: Wheelchair Skills Training - In Person

INTERVENTIONS:
Behavioral: Wheelchair Skills Training - Remote — Individuals will receive wheelchair skills training remotely. They will be provided with the Wheelchair Skills Training Program to review (http://www.wheelchairskillsprogram.ca/eng/index.php), and then will be directed to use this information to perform the wheelchair skills. They will video the attempts, and will receive feedback on methods to improve their techniques.
  Arms: Wheelchair Skills Trainers
Behavioral: Wheelchair Skills Training - In Person — Individuals will receive wheelchair skills training in one-on-one sessions, taught by those who received the wheelchair skills training remotely.
  Arms: Wheelchair Skills Trainees

SUMMARY:
The objective of the study is to evaluate the effectiveness of remote training to teach clinicians how to train others in wheelchair skills.

ELIGIBILITY:
Inclusion Criteria:

• Age 18 to 75

Exclusion Criteria:

• Upper or lower extremity injury that would preclude the ability to use a wheelchair.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in wheelchair skills capacity of trainees at study completion as measured by the Wheelchair Skills Test Questionnaire | Baseline, and at study completion ( an average of 3 weeks)
  Trainees will have increased capacity to perform wheelchair skills after receiving one-on-one skills training.
Change from baseline in wheelchair skills confidence of trainees at study completion as measured by the Wheelchair Skills Test Questionnaire | Baseline, and at study completion ( an average of 3 weeks)
  Trainees will have increased confidence in their ability to perform wheelchair skills after receiving one-on-one skills training.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boninger, M.D., Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - South Florida Spinal Cord Injury System, Miami, Florida
  - Midwest Regional Spinal Cord Injury Care System, Chicago, Illinois
  - Northern New Jersey Spinal Cord System, West Orange, New Jersey
  - University of Pittsburgh Model Center on Spinal Cord Injury, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD outside of collaborators.

REFERENCES:
- [Derived] Worobey LA, Kirby RL, Cowan RE, Dyson-Hudson TA, Shea M, Heinemann AW, Pedersen JP, Boninger ML. Efficacy of a Remote Train-the-Trainer Model for Wheelchair Skills Training Administered by Clinicians: A Cohort Study With Pre- vs Posttraining Comparisons. Arch Phys Med Rehabil. 2022 Apr;103(4):798-806. doi: 10.1016/j.apmr.2021.03.042. Epub 2021 Jun 6. PMID 34090853

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT03499951/Prot_SAP_000.pdf